CLINICAL TRIAL: NCT00883233
Title: Efficacy and Safety Comparison of Four Different Regimens of Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel in the Treatment of Acne Vulgaris
Brief Title: Comparison of Four Different Regimens of Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel in Acne Vulgaris
Acronym: FREE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Jean-Charles DHUIN Clinical Trial Manager, Galderma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29085
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2010-11

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel 3-hour daily application before bedtime for first 4 weeks and then standard overnight daily application for the following 8 weeks
  Interventions: Drug: Adapalene-BPO 3-hour daily application before bedtime
- 2 (Experimental): Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel every other day application for the first 4 weeks and then standard overnight daily application for the following 8 weeks
  Interventions: Drug: Adapalene-BPO Gel every other day application
- 3 (Experimental): Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel standard daily overnight application with Cetaphil® Moisturizing Lotion application at wake-up time for the first 4 weeks and then standard daily overnight application for the following 8 weeks
  Interventions: Drug: Adapalene-BPO Gel standard+Cetaphil® Moisturizing Lotion
- 4 (Active Comparator): Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel standard daily overnight application for 12 week
  Interventions: Drug: Adapalene BPO Gel standard daily overnight application

INTERVENTIONS:
Drug: Adapalene BPO Gel standard daily overnight application — Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel standard daily overnight application for 12 week
  Other Names: Standard
  Arms: 4
Drug: Adapalene-BPO 3-hour daily application before bedtime — Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel 3-hour daily application before bedtime for first 4 weeks and then standard overnight daily application for the following 8 weeks
  Other Names: 3-hour before bedtime
  Arms: 1
Drug: Adapalene-BPO Gel every other day application — Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel every other day application for the first 4 weeks and then standard overnight daily application for the following 8 weeks
  Other Names: every other day
  Arms: 2
Drug: Adapalene-BPO Gel standard+Cetaphil® Moisturizing Lotion — Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel standard daily overnight application with Cetaphil® Moisturizing Lotion application at wake-up time for the first 4 weeks and then standard daily overnight application for the following 8 weeks
  Other Names: Adapalene-BPO Gel with Cetaphil® Moisturizing Lotion
  Arms: 3

SUMMARY:
The purpose of this study is to compare the tolerability of 3 treatment regimens containing Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel with that of Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel standard daily overnight application for 12 weeks in the treatment of acne vulgaris. The efficacy of the four treatment regimens will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Subjects of any race, aged 12 to 35 years inclusive
* Subjects with mild or moderate facial acne vulgaris
* Subjects with skin phototype I to IV

Exclusion Criteria:

* Subjects with more than 1 nodules or cysts on the face,
* Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.)

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Tan, MD, Principal Investigator — Windsor, ON, Canada
Locations (2):
- Canada (2):
  - Galderma Investigational Site, Windsor, Ontario
  - Galderma Investigational Site, Montreal, Quebec

REFERENCES:
- See also: Related Info — http://www.galderma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 23 APR 2009 to 09 SEP 2009 in three private practice Canadian centres. Two centers used a central IRB, and the other used a local IRB.
Groups:
- Adapalene-BPO Gel 3h: Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel 3-hour daily application before bedtime for first 4 weeks and then standard overnight daily application for the following 8 weeks
- Adapalene-BPO Gel EoD: Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel every other day application for the first 4 weeks and then standard overnight daily application for the following 8 weeks
- Adapalene-BPO Gel Cetaphil: Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel standard daily overnight application with Cetaphil® Moisturizing Lotion application at wake-up time for the first 4 weeks and then standard daily overnight application for the following 8 weeks
- Adapalene-BPO Gel StD: Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel standard daily overnight application for 12 week
Period: Overall Study
Arm/Group | Adapalene-BPO Gel 3h | Adapalene-BPO Gel EoD | Adapalene-BPO Gel Cetaphil | Adapalene-BPO Gel StD
Started | 32 | 32 | 29 | 30
Completed | 27 | 28 | 25 | 25
Not Completed | 5 | 4 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene-BPO Gel 3h | Adapalene-BPO Gel EoD | Adapalene-BPO Gel Cetaphil | Adapalene-BPO Gel StD | Total
Number analyzed (Participants) | 32 | 32 | 29 | 30 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 13 | 14 | 57
  Between 18 and 65 years | 17 | 17 | 16 | 16 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (6.5) | 20.4 (6.39) | 20.9 (6.83) | 20.8 (6.31) | 20.6 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 16 | 16 | 71
  Male | 12 | 13 | 13 | 14 | 52
Region of Enrollment [Number; unit: participants]
  Canada | 32 | 32 | 29 | 30 | 123

OUTCOME MEASURES:

1. Primary Outcome: Local Tolerability Was Analyzed in Terms of Worst Score Post-Baseline.
Description: Total Sum Score (TSS) is the sum of the 4 local tolerability scores for dryness, erythema, scaling and stinging/burning evaluated at each visit [None=0, Mild=1, Moderate=2 and Severe=3]. In consequence, it ranges from 0 [better outcome] to 12 [worse outcome]and was calculated for each study visit.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Adapalene-BPO Gel 3h | Adapalene-BPO Gel EoD | Adapalene-BPO Gel Cetaphil | Adapalene-BPO Gel StD
Number analyzed (Participants) | 32 | 32 | 29 | 30
Scores on a scale | 4.23 (2.04) | 3.06 (1.92) | 3.25 (2.05) | 4.13 (2.45)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Adapalene-BPO Gel 3h | Adapalene-BPO Gel EoD | Adapalene-BPO Gel Cetaphil | Adapalene-BPO Gel StD
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 8/32 | 5/32 | 8/29 | 6/30
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene-BPO Gel 3h (N=32) | Adapalene-BPO Gel EoD (N=32) | Adapalene-BPO Gel Cetaphil (N=29) | Adapalene-BPO Gel StD (N=30)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
sunburn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
upper track respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
skin oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor for review and approval at least 2 months prior to the date of the intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.